CLINICAL TRIAL: NCT04157556
Title: The Effect of Maximal Exercise on Matrix Metalloproteinase Enzyme and Its Inhibitor (MMP9 and TIMP1) and The Role of MMP9 -1562 C/T and TIMP1 372 T/C Polymorphisms
Brief Title: The Effect of Maximal Exercise on MMP9 and TIMP1 and The Role of MMP9 -1562 C/T and TIMP1 372 T/C Polymorphisms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Collaborators: Ege University (Other)
Responsible Party: Principal Investigator, Merve Koca Kosova, research assistant, Dokuz Eylul University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18-7.1/49
Record Dates: First submitted 2019-11-05; First posted 2019-11-08 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: MMP9; TIMP1; MMP9 -1562 C/T; TIMP1 372 T/C

STUDY DESIGN:
Intervention Model Description: There are 2 groups in the study: Athletes and sedentary people.They will apply the same acute exercise protocol (The Yo-Yo Intermittent Recovery Test Level 1). A blood test will conduct before and after the acute exercise protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group of athletes (Experimental): Age: 18-35 Gender: Male Basketball, volleyball, handball players who have been training regularly for at least last 3 months.
  Interventions: Other: Yo-Yo Intermittent Recovery Test Level 1
- Group of sedentary people (Experimental): Age: 18-35 Gender: Male Individuals with similar physical characteristics to the group of athletes and who have not exercise regularly for at least last 3 months.
  Interventions: Other: Yo-Yo Intermittent Recovery Test Level 1

INTERVENTIONS:
Other: Yo-Yo Intermittent Recovery Test Level 1 — The test is a standard test battery with progressively increasing speeds. After every 40-m run (2x20 m), active rest is performed by walking or jogging at a distance of 10 m (2x5 m). for 10 seconds. Participants are trying to adjust their speed according to incoming audio signals.The test is terminated when the participants can not reach the signal twice. The test ends in 10-20 minutes depending on the level of participants.
  Reference Bangsbo, J., Iaia, F. M., & Krustrup, P. (2008). The Yo-Yo intermittent recovery test. Sports medicine, 38(1), 37-51.
  Krustrup, P., Mohr, M., Amstrup, T., Rysgaard, T., Johansen, J., Steensberg, A., ... & Bangsbo, J. (2003). The yo-yo intermittent recovery test: physiological response, reliability, and validity. Medicine & Science in Sports & Exercise, 35(4), 697-705.

SUMMARY:
Matrix metalloproteinases (MMPs) play a critical role in the remodeling and regeneration of skeletal muscle. Studies which investigate exercise and effects of MMPs and tissue inhibitors of matrix metalloproteinases (TIMPs) are contradictory. Also the role of MMP9 -1562 C/T and TIMP1 372 T/C polymorphisms on exercise are unclear. In accordance with this conditions the hypothesis of the study are as follows:

1. Levels of basal serum MMP9 and TIMP1 are different between athletes (volleyball, basketball, handball) and sedentary people.
2. Levels of serum MMP9 and TIMP1 response to maximal exercise are different between athletes (volleyball, basketball, handball) and sedentary people .
3. Relationship between levels of serum MMP9 and TIMP1 response to maximal exercise are different between athletes (volleyball, basketball, handball) and sedentary people.
4. Levels of basal serum MMP9 and TIMP1 are related to MMP9 -1562 C/T and TIMP1 372 T/C polymorphisms.
5. Relationship between levels of serum MMP9 and TIMP1 response to maximal exercise and MMP9 -1562 C/T and TIMP1 372 T/C polymorphisms are different between athletes (volleyball, basketball, handball) and sedentary people.

ELIGIBILITY:
Inclusion Criteria:

Group of athletes:

* Male basketball players who have been training regularly for at least last 3 months.
* Male volleyball players who have been training regularly for at least last 3 months.
* Male handball players who have been training regularly for at least last 3 months.

Group of sedentary people:

* Male individuals with similar physical characteristics to the group of athletes
* Male individuals who have not exercise regularly for at least last 3 months.

Exclusion Criteria(For two groups):

* Smoking regularly
* Drinking alcohol regularly
* Using drug and antioxidant substance
* Being obese,
* Being sick or having disability

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-01-03 (Actual); Study Completion 2020-04-28 (Actual)

PRIMARY OUTCOMES:
Level of MMP9 and TIMP1 | Yo-Yo Intermittent Recovery Test level 1 (the test performed until the subject is exhausted, the test lasts 10-20 minutes according to endurance capacity of the participants)
  The effect of acute maximal exercise on serum MMP9 and TIMP1 levels in athletes and sedentary people.
MMP9 -1562 C/T, TIMP1 372 T/C polymorphisms | Yo-Yo Intermittent Recovery Test level 1 (the test performed until the subject is exhausted, the test lasts 10-20 minutes according to endurance capacity of the participants)
  The role of MMP9 -1562 C/T and TIMP1 372 T/C polymorphisms on the effect of acute maximal exercise on serum MMP9 and TIMP1 in athletes and sedentary people.

SECONDARY OUTCOMES:
Level of indicators of muscle damage and inflammation and oxidative stress | Yo-Yo Intermittent Recovery Test level 1 (the test performed until the subject is exhausted, the test lasts 10-20 minutes according to endurance capacity of the participants)
  The relationship between primary outcome measures and indicators of muscle damage, inflammation and oxidative stress.
  Indicators to be determined: creatine kinase (CK), aspartate aminotransferase (AST), alanine aminotransferase (ALT), Interleukin-6 (IL-6), C- reactive protein (CRP), total antioxidant status (TAS), total oxidant status (TOS), nitric oxide (NO)
Level of blood lipids and lipoproteins, glucose, urea, creatinine, hemogram | Yo-Yo Intermittent Recovery Test level 1 (the test performed until the subject is exhausted, the test lasts 10-20 minutes according to endurance capacity of the participants)
  The relationship between primary outcome measures and blood lipids and lipoproteins, glucose, urea, creatinine and hemogram

CONTACTS AND LOCATIONS:
Overall Officials: Faruk Turgay, associate professor, Study Chair — Ege University, Faculty of Sports Science
Locations (1):
- Ege University Faculty of Sports Science, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided